CLINICAL TRIAL: NCT06845930
Title: Rectal Versus Intramuscular Diclofenac for Pain Relief Following Elective Caesarean Section at Alex Ekwueme Federal University Teaching Hospital Abakaliki: A Randomized Controlled Trial
Brief Title: Rectal Versus Intramuscular Diclofenac for Pain Relief Following Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assumpta Nnenna Nweke (Other Government)
Responsible Party: Sponsor-Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Organization: Federal Teaching Hospital Abakaliki (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AEFUTHA/REC/VOL 3/2020/038
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Painrelief; Postoperative
Keywords: Rectal diclofenac; Caesarean section

STUDY DESIGN:
Intervention Model Description: open label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal diclofenac (Experimental): Participants had 100mg of rectal diclofenac administered immediately after skin closure by the researcher. The medication was repeated every 12hourly for 24 hours. For all the participants, 30 mg pentazocine was given intramuscularly every 6 hours for 24 hours.
  Interventions: Drug: Rectal Diclofenac
- Intramuscular diclofenac (Active Comparator): Participants had 75mg of intramuscular diclofenac administered immediately after skin closure by the researcher. The medication was repeated every 12hourly for 24 hours. For all the participants, 30 mg pentazocine was given intramuscularly every 6 hours for 24 hours.
  Interventions: Drug: Intramuscular diclofenac

INTERVENTIONS:
Drug: Rectal Diclofenac — Rectal diclofenac, 100mg administered immediately after skin closure then 12 hourly for 24 hours.
  Arms: Rectal diclofenac
Drug: Intramuscular diclofenac — Intramuscular diclofenac, 7mg administered immediately after skin closure then 12 hourly for 24 hours.
  Arms: Intramuscular diclofenac

SUMMARY:
Caesarean section (CS) is one of the commonest major Obstetric surgeries worldwide and its rate has markedly increased globally. Pain control is an integral part of enhancement of recovery after caesarean section and NSAIDs have been used in combination with opioids for post-operative pain management in recent times. There are sparse data on maternal satisfaction with suppository diclofenac or any data from our centre that compared the intramuscular and rectal routes of diclofenac administration. Hence this study was conceived to compare the efficacy of rectal diclofenac and intramuscular diclofenac as an adjunct to intramuscular pentazocine in the management of post-operative pain in women who have elective caesarean section.

DETAILED DESCRIPTION:
Background: Caesarean section (CS) is one of the commonest major Obstetric surgeries worldwide and its rate has markedly increased globally. Pain control is an integral part of enhancement of recovery after caesarean section and NSAIDs have been used in combination with opioids for post-operative pain management in recent times. There are sparse data on maternal satisfaction with suppository diclofenac or any data from our centre that compared the intramuscular and rectal routes of diclofenac administration. Hence this study was conceived to compare the efficacy of rectal diclofenac and intramuscular diclofenac as an adjunct to intramuscular pentazocine in the management of post-operative pain in women who have elective caesarean section.

Aim: This study is designed to compare the efficacy of rectal diclofenac with that of intramuscular diclofenac as pain relief among women after elective Caesarean section at Alex-Ekwueme Federal University Teaching Hospital, Abakaliki.

Methods: This was a randomized equivalence controlled trial conducted among pregnant women booked for elective Caesarean section at Alex-Ekwueme Federal University Teaching Hospital Abakaliki, comparing the efficacy of rectal diclofenac with that of intramuscular diclofenac as pain relief among women after elective caesarean section at term. One arm received 100mg of suppository diclofenac and the other arm received 75mg of intramuscular diclofenac. These doses were repeated every 12hours for 24 hours. Pain scoring was done at 1, 6, 12, 18 and 24 hours after administration of the drugs. The data obtained was analysed using IBM SPSS software (version 23, Chicago II, USA) and the intention to treat concept. A difference with a P value of ≤ 0.05 was taken to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section at term with spinal anaesthesia;E

Exclusion Criteria:

1. Allergy to NSAIDS
2. Bleeding diathesis
3. Use of general anesthesia
4. Chronic liver disease
5. History of renal disease
6. Asthma in pregnancy
7. Emergency Cesarean section
8. Morbid obesity
9. Sickle cell anaemia patients
10. Hypertensive disorders of pregnancy
11. Refusal to give consent

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post caesarean section
Enrollment: 60 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Pain score after the administration of the rectal and intramuscular diclofenac | 24 hours after the last dose
  Pain score at different intervals with either rectal or intramuscular diclofenac immediately after skin closure. This pain assessment was done with visual analogue scale ranging from 0 to 10. zero represents no pai while ten represents the worst possible pain.

SECONDARY OUTCOMES:
maternal side effects and need for additional analgesia | 24 hours after the last dose
  Number of participants with local irritation at the site of injection or insertion of drug,headache,dizziness and loss of appetite. a Also the number of participants requiring additional analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No